CLINICAL TRIAL: NCT01469702
Title: Open Label Study of Prednisone and Azithromycin in the Treatment of Patients With Cat Scratch Disease
Brief Title: The Efficacy of Prednisone and Azithromycin in the Treatment of Patients With Cat Scratch Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, director R&D devision, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-11-MG-0232-11-TLV-CTIL
Record Dates: First submitted 2011-09-13; First posted 2011-11-10 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Cat-scratch Disease; Bartonella Infections
Keywords: cat-scratch disease; Bartonella henselae; corticosteroids; treatment
MeSH Terms: conditions — Cat-Scratch Disease; Bartonella Infections | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: prednison and azithromycin — Patients with typical cat-scratch disease will be treated with a 5-day course of prednison and azithromycin.
Drug: prednison, azithromycin — Cap Azithromycin 500 mg qd (first day), then 250 mg qd for 4 days and Tab prednison 1 mg/kg/day, not exceeding 60 mg/day, qd, for 5 days.
Drug: prednison, Azenil — Cap Azenil 500 mg qd (first day), then 250 mg qd for 4 days and Tab prednison 1 mg/kg/day, not exceeding 60 mg/day qd, for 5 days.

SUMMARY:
Bartonella henselae is the etiologic agent of cat scratch disease (CSD). 90% of patients present with regional lymphadenitis (typical CSD) while 10% will have disease involving other organs, such as neuroretinitis, arthropathy, erythema nodosum, and encephalitis (atypical CSD). In most CSD cases resolution occurs in 2 to 3 months although a prolonged course often occurs. Data on the efficacy of antibiotic therapy in CSD is limited. Azithromycin has been shown to have a small favorable effect in a small comparative study and is commonly prescribed for CSD, however its overall effect is not satisfactory. Corticosteroids may be effective in the treatment of CSD for the following reasons:

* Many experts believe that host response is involved in the pathogenesis of CSD and is responsible for the clinical manifestations rather than the direct effect of B. henselae. The absence of viable organisms in affected lymph nodes (in the presence of positive PCR for B. henselae DNA), and the fact that arthritis, arthralgia and erythema nodosum (that are often associated with autoimmune diseases) have been described in CSD, support this concept.
* Corticosteroids have been anecdotally reported to have been administered to patients with CSD, apparently with some success. The purpose of this study is to evaluate the efficacy of corticosteroids in addition to azithromycin in CSD. The study hypothesis is that corticosteroids will improve out come. Ten patients with typical CSD will be treated with a 5-day oral course of prednisone (1 mg/kg up to 60 mg/day) and azithromycin (500 mg on day 1 and 250 mg on days 2-5). Patients will be under followed up for 3 months. Major outcome measures will include duration of symptoms and signs, with particular emphasis on affected lymph node size and duration using a specific scoring system (lymphadenitis score, LS). LS will be used to evaluate lymphadenitis at each follow-up visit. The time period from baseline LS until 75% and 90% reduction in LS in the treatment group will be compared with historical controls. The historical control group will be consisted of age, sex, and clinical manifestations-matched CSD patients who were treated with azithromycin without corticosteroids.

ELIGIBILITY:
Inclusion criteria

* Patients and/or legally authorized representative(s), if applicable, who have been fully informed and have given voluntary written informed consent OR patients unable to write and/or read but who fully understand the oral information given by the Investigator (or nominated representative) who have given oral informed consent witnessed in writing by an independent person.
* Ability and willingness to comply with the protocol.
* Male and female patients aged 14-60 years at the time of signing informed consent.
* Female patients must be non-lactating and at no risk of pregnancy for one of the following reasons: Postmenopausal (amenorrhea for at least 1 year); post hysterectomy and/or post-bilateral ovariectomy; if of childbearing potential, having a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test at screening and is using a highly effective method of birth control throughout the study; reliable sexual abstinence throughout the course of the study is acceptable as a highly effective method of birth control for the purposes of this study.
* Patients with clinical manifestations consistent with early typical cat scratch disease (lymphadenitis) before spontaneous improvement has been recorded and before development of suppuration.
* Laboratory confirmation (serology and/or PCR) of cat scratch disease

Exclusion criteria

* Women who are pregnant or breastfeeding.
* Known history of allergy, hypersensitivity, or any serious reaction to azithromycin, other macrolides or corticosteroids.
* Patients for whom azithromycin or corticosteroids is contra-indicated.
* Patients at high risk for QT/QTc prolongation, e.g. Baseline prolongation of QTcF >/=500 msec; Risk factors for Torsade de Pointes (e.g. uncompensated heart failure, abnormal potassium or magnesium levels that cannot be corrected, any unstable cardiac condition during the last 30 days, or a family history of long QT syndrome); The use of concomitant medications that prolong the QT/QTc interval.
* Current treatment with systemic corticosteroids.
* Patients with typical late cat scratch disease who has demonstrated constant improvement in the clinical manifestations of the involved lymph node.
* Atypical cat scratch disease (e.g. encephalitis, pneumonitis, osteomyelitis).
* Endocarditis due to Bartonella sp..
* Diabetes mellitus.
* Peptic ulcer disease or history of upper GI bleeding.
* History of inadequately treated tuberculosis or evidence of tuberculosis in the chest radiography.
* Schizoaffective disorder, anxiety or depression treated with antipsychiatric drugs, at present or in the past.
* AIDS or positive serology for HIV.
* Absolute neutrophil count < 1000/mm3.
* Treatment with any investigational drug in any clinical trial within 30 days prior to administration of study medication.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Severity score of lymphadenitis using a lymphadenitis Score (LS). | Change from baseline in LS until 75% and 90% reduction in LS
  LS will evaluate the severity of lymphadenitis, using the following clinical parameters: size of lymph node in cm; pain estimated by the patient, using a 0-5 scale (0 equals no pain, 5 the most severe pain); tenderness estimated by the physician, (0 equals no tenderness, 5 the most severe tenderness); erythema of the skin overlying the affected lymph-node (0 no erythema, 1 mild erythema, 2 moderate erythema and 3 severe erythema); suppuration of a lymph node will score 5 points, no suppuration will score 0. The total score will consist of the arithmetical summation of the 5 parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- The Infectious Disease Unit, Tel Aviv Medical Center, Tel Aviv, Israel